CLINICAL TRIAL: NCT07402122
Title: Development and Implementation of a Transparent Registry Based on FAIR Principles for Duchenne and Becker Muscular Dystrophy (DBMD) Under the Auspices of the Society for Neuropediatrics (GNP) - FAIR-DMD
Brief Title: Registry for Duchenne and Becker Muscular Dystrophy
Acronym: FAIR-DMD
Status: Not yet recruiting | Type: Observational
Sponsor: Dr. Andreas Ziegler (Other)
Responsible Party: Sponsor-Investigator, Dr. Andreas Ziegler, Head of paedKliPS (Pediatric Clinical Pharmacology Study Center), University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Other Study IDs: 25-12847-BO
Record Dates: First submitted 2026-01-16; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Duchenne Muscular Dystrophy (DMD); Becker Muscular Dystrophy; Dystrophinopathy Symptomatic Female Carrier
Keywords: Muscular Dystrophies; Duchenne Muscular Dystrophy; Becker Muscular Dystrophy; Muscular Dystrophy; Dystrophinopathy; FAIR Principles; Neuromuscular Diseases; Health Related Quality of Life (HRQoL)
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Duchenne muscular dystrophy (DMD) is an X-linked, recessive, progressive, and degenerative neuromuscular disorder that affects approximately one in 5,000 newborn boys. The established "standard of care" has improved prognosis; however, a causal therapy is not yet available. In 2024 and 2025, the first disease-modifying therapies were approved. These include Vamorolone (Agamree®) as a corticosteroid replacement with a more favorable side-effect profile for children aged four and older, and Givinostat (Duvyzat®) as a combination therapy with corticosteroids for ambulatory boys aged six and older. In this context, the FAIR-DMD Registry was initiated. The registry is based on the so-called FAIR principles. The acronym FAIR stands for the data principles Findable, Accessible, Interoperable and Reusable. The international FAIR principles are guidelines for the description, storage, and publication of scientific or administrative data. The FAIR-DMD registry is a disease-specific, academically managed registry for patients with Duchenne and Becker muscular dystrophy (DMD/BMD). Its goal is to systematically collect clinical data, scientifically monitor new disease-modifying therapies in routine care, and create an evidence-based foundation for the further development of diagnostics, therapy, and care structures. Furthermore, the registry collects data on patients' health related quality of live using an app for data entry. The FAIR-DMD Registry is being established under the auspices of the Society for Neuropediatrics (GNP) and operated in close coordination with Swiss Registry for Neuromuscular Disorders (Swiss-Reg-NMD). The GNP is a non-profit professional society that covers the entire spectrum of neuropediatric topics in clinical and cross-sector care. In the planned pilot phase, the GNP will act as trustee for financing. This model creates the opportunity to structurally address central challenges in health services research and establish a high-quality, internationally compatible registry structure. In the long term, the FAIR-DMD Registry aims to significantly improve care for DMD and BMD patients in German-speaking countries, evaluate the effectiveness of new therapies in clinical practice, and establish binding frameworks for quality-assured care.

DETAILED DESCRIPTION:
The FAIR-DMD registry is a disease-specific, academically managed registry for patients with Duchenne and Becker muscular dystrophy (DMD/BMD).

Already in early childhood, affected boys show nonspecific developmental abnormalities, such as delays in speech or cognitive development or delayed achievement of motor milestones. Diagnosis is usually made between the ages of three and five through markedly elevated creatine kinase (CK) levels and molecular genetic analyses. The disease course is progressive: after a plateau phase in the preschool years, increasing muscle weakness-despite corticosteroid therapy-typically leads to loss of ambulation in early adolescence. Secondary complications arise from cardiac and respiratory involvement. Life-limiting factors include progressive cardiomyopathy, cardiac arrhythmias, and global respiratory failure, which usually necessitates non-invasive ventilation in early adulthood.

Currently, 26 specialized treatment centers in Germany and 5 in Austria are participating in the project. In Switzerland, a registry for DBMD patients is already being maintained, the Swiss Registry for Neuromuscular Disorders (Swiss-Reg-NMD). The registry is open to all centers that wish to participate in the future. Within the FAIR-DMD project, interoperability between FAIR-DMD and the Swiss registry is being pursued, and additional disease-specific and academically managed European Duchenne registries could be further developed for future data exchange. Data from patients treated with new disease-modifying therapies - which may in the future alter the progression of DMD and BMD - will also be included in the project.

Aims of the study are:

* Harmonization and standardization of care
* Support and evaluation of new disease-modifying therapies
* Improvement of care quality
* Establishment of the registry as an independent research tool
* Ensuring international cooperation and comparability
* Patient-centered approach and collection of subjective indicators
* Aim for sustainability and implementation into routine care To achieve these aims apart of the registry a telemedicine platform will be implemented. The telemedicine platform consists of a web-based dashboard for study personnel and an app for patients. The app will be used for appointment management, communication with the treating doctor and health care professionals, and to fill out Health Related Quality of Life questionnaires. Data from the telemedicine platform will automatically be transferred to the registry and vice versa.

Another measure in the FAIR-DMD project is to simplify the management of adverse drug reactions (ADR). New therapies are often approved despite very small patient populations in clinical trials. As a result, the majority of knowledge regarding their benefits - but especially their potential risks - emerges only after approval. In the future, as soon as new ADRs occur, they must be managed as effectively as possible, drawing on all available expertise and experience, following a "best practice" approach. Alongside the existing legally mandated ADR reporting procedures to the federal authorities and pharmaceutical companies, the process of digitally supported documentation of the clinical course following the occurrence of an ADR is to be optimized.

In FAIR-DMD it is planned that the report of an occurring ADR shall be automatically forwarded to the relevant authorities through the telemedicine platform, without requiring the same forms to be completed multiple times. To achieve this, we work very closely with the federal authority and pharmaceutical companies.

In addition to these measures FAIR-DMD aims to establish a therapy recommendation board, which also uses the telemedicine platform.

Our mission is to harmonize and standardize care for patients with dystrophinopathies, ensuring high-quality treatment and equitable access. We aim to support and evaluate innovative disease-modifying therapies, establish the registry as an independent research instrument, and foster international collaboration for global comparability. By prioritizing patient-centered approaches and integrating subjective indicators, we strive for sustainability and seamless implementation into routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed diagnosis of dystrophinopathy
* Female carriers only if they show clinical symptoms of a dystrophinopathy
* Treatment in one of the participating centers
* No age restrictions
* Ability to understand the patient information and sign the informed consent
* Consent capability by the patient themselves and/or by the parents
* Agreement to data exchange between the treating physicians, the telemedicine platform, and the registry
* Possession of a tablet or a smartphone

Exclusion Criteria:

* Missing legally valid consent form from the patient and/or legal guardians
* Project content is not understandable to the participant and/or legal guardians
* Not in possession of a tablet or smartphone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients meeting the eligibilty criteria in Germany and Austria.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2040-12 (Estimated); Study Completion 2041-06 (Estimated)

PRIMARY OUTCOMES:
EQ-5D-5L | * "Baseline" * "every six months" * "through study completion, maximum 15 years"
  The EQ-5D is a validated generic instrument for measuring health-related quality of life. It assesses five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and enables the calculation of a health index from 0 (very poor) to 1 (best possible health).
EQ VAS | * "Baseline" * "every six months" * "through study completion, maximum 15 years"
  A visual analog scale on which patients rate their current state of health on a scale from 0 ("worst possible") to 100 ("best possible").
DMD-QoL | * "Baseline" * "every six months" * "through study completion, maximum 15 years"
  The DMD-QoL is a disease-specific questionnaire designed to assess the health-related quality of life of people with Duchenne muscular dystrophy. It takes into account physical, emotional, and social aspects as well as the impact of the disease on everyday life. In the DMD-QoL, the raw values of the individual scales are usually transformed onto a scale from 0 to 100. 0 represents the worst possible health-related quality of life, while 100 represents the best possible health-related quality of life-higher values therefore indicate a better perceived quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Schara-Schmidt, Prof. Dr., Principal Investigator — Universitätsklinikum Essen, Klinik für Kinderheilkunde; Andreas Ziegler, Dr., Study Director — Universitätsklinikum Heidelberg, Zentrum für Kinder- und Jugendmedizin
Locations (2):
- Germany (2):
  - Universitätsklinikum Essen Klinik für Kinderheilkunde I, Essen
  - Universitätsklinik Heidelberg, Zentrum für Kinder- und Jugendmedizin, Heidelberg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: App used in the study. — https://www.one4app.com/